CLINICAL TRIAL: NCT05456919
Title: Quality of Sexual Function in BRCA Mutated Women
Acronym: BRCA_SFQ28
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Federico Ferrari, Research Associate, Università degli Studi di Brescia
Other Study IDs: BRCA_SFQ28
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: BRCA Mutation; Sexual Dysfunction; Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological
Keywords: brca; sexual
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Coitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BRCA Mutated and no RRS
  Interventions: Other: SFQ28 Questionnaire
- BRCA Mutated and RRS
  Interventions: Other: SFQ28 Questionnaire
- BRCA Mutated and oncological diagnosis
  Interventions: Other: SFQ28 Questionnaire
- BRCA Wildtype without oncological diagnosis
  Interventions: Other: SFQ28 Questionnaire

INTERVENTIONS:
Other: SFQ28 Questionnaire — SFQ28 Questionnaire

SUMMARY:
Quality of sexual function in BRCA mutated women is investigated using SFQ28 questionnaire.

DETAILED DESCRIPTION:
We aim to investigate and compare the impact of diagnosis of BRCA, the impact of risk reducing surgery (RRS) and oncological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* TBC

Exclusion Criteria:

* TBC

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: TBC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of SFQ28 Score | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Federico Ferrari, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No